CLINICAL TRIAL: NCT05287984
Title: A Phase 2 Clinical Trial to Evaluate the Efficacy of Zanubrutinib Followed Zanubrutinib Plus FCR (Fludarabine Cyclophosphamide and Rituximab) / BR(Bendamustine and Rituximab) in Newly Diagnosed Symptomatic CLL/SLL (STOP Trial)
Brief Title: Zanubrutinib Followed Zanubrutinib Plus FCR / BR in Newly Diagnosed Symptomatic CLL/SLL
Acronym: ZFCR/ZBR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Yi Shuhua, Professor, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BDH-CLL-002-2022/02/14
Record Dates: First submitted 2022-02-26; First posted 2022-03-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Newly Diagnosed
Keywords: chronic lymphocytic leukemia; Small Lymphocytic Lymphoma; newly diagnosed; Zanubrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; fludarabine; Cyclophosphamide; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZFCR regimen (Experimental): Patients aged 65 years or younger who can tolerate FCR： Patients in this group will receive zanubrutinib monotherapy for 12 months, then receive 4 cycles of zanubrutinib, fludarabine, cyclophosphamide and rituximab(ZFCR). Efficacy evaluation and MRD test of peripheral blood and bone marrow were performed at the 17th cycle after 16 cycles to obtain study end point data. Patients with CR/CRi and MRD negative could stop taking zanubrutinib, and other patients could stop taking zanubrutinib or continue treatment. Follow-up and efficacy assessment were conducted every three months.
  Interventions: Drug: Zanubrutinib, Fludarabine, cyclophosphamide and rituximab
- ZBR regimen (Experimental): For patients older than 65 years or who cannot tolerate FCR regimens: Patients in this group will receive zanubrutinib monotherapy for 12 months, then receive 4 cycles of bendamostine and rituximab(BR). Efficacy evaluation and MRD test of peripheral blood and bone marrow were performed at the 17th cycle after 16 cycles to obtain study end point data. Patients with CR/CRi and MRD negative could stop taking zanubrutinib and other patients could stop taking zanubrutinib or continue treatment.
  Interventions: Drug: Zanubrutinib, bendamustine, rituximab

INTERVENTIONS:
Drug: Zanubrutinib, Fludarabine, cyclophosphamide and rituximab — Patients aged 65 years or younger who can tolerate FCR.
  Other Names: ZFCR regimen
  Arms: ZFCR regimen
Drug: Zanubrutinib, bendamustine, rituximab — For patients older than 65 years or who cannot tolerate FCR regimens.
  Other Names: ZBR regimen
  Arms: ZBR regimen

SUMMARY:
This study aims to evaluate the long-term efficacy of BTK inhibitor Zanubrutinib monotherapy , sequential Zanubrutinib combined (Fludarabine, cyclophosphamide and rituximab /bendamustine and rituximab)FCR/BR regimen by a limited period of treatment for the newly diagnosed Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL). The investigators propose this combination will improve the MRD negative rate of patients with CR/CRi after treatment was significantly higher than that of FCR chemotherapy can be a time-limited regimen which will reduce the life-time therapy and benefit the patients.

DETAILED DESCRIPTION:
The investigators designed timed FCR/BR treatment for BTK inhibitor Zanubrutinib monotherapy after continuous remission, which shortened the treatment time, deepened the depth of remission, and enabled some patients to achieve deep remission (MRD negative), and realized long-term survival after drug withdrawal. Treatment regimens: Zanubrutinib monotherapy for 12 months followed by 4 courses of immunochemotherapy with FCR or BR. Cohort 1 was designed to apply FCR for patients aged 65 years or younger who could tolerate FCR. Cohort 2 was designed to apply BR in patients older than 65 years or unable to tolerate FCR.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 Years and older (Adult, Older Adult)
* 2. Age >65 years or age ≤65 years with creatinine clearance of 30-69 mL/min or patients with a cumulative Disease Rating Scale (CIRS-G) score greater than 6 point were enrolled in cohort 2 , other patients were enrolled in cohort 1.
* 3. Confirmed diagnosis of CLL or SLL that meets the 2008 IWCLL criteria
* 4. The patients are untreated or without prior systemic therapy for disease, the specific conditions are as follows:
* a) Prior treatment with a fludarabine or treatment with bendamustine or rituximab regimen
* b) Not treated with Chlorambucil, or treated with Chlorambucil for less than 4 weeks (alone or in combination with adrenal glucocorticoid)
* c) If the above treatment has been applied, it is necessary to stop treatment for 2 weeks before joining the group for treatment
* 5. Treatment indications for CLL mainly include (meeting at least one of the following conditions):
* a) Evidence of progressive bone marrow failure presenting as progressive decrease in hemoglobin and/or platelets
* b) Splenomegaly (e.g., >6cm below the left costal margin) or progressive or symptomatic splenomegaly
* c) giant lymph node enlargement (longest diameter >10cm) or progressive or symptomatic lymph node enlargement
* d) Progressive lymphocytosis, such as lymphocytosis >50% within 2 months, or lymphocyte multiplication time (LDT) <6 months. When the initial lymphocyte was <30×109/L, LDT alone could not be used as a treatment indication
* e) Autoimmune hemolytic anemia (AIHA) and/or immune thrombocytopenia (ITP) do not respond well to corticosteroids or other standard treatments
* f) Symptoms associated with at least one of the following diseases: ①≥10% weight loss with no apparent cause in the previous 6 months; ② Severe fatigue (such as ECOG physical state ≥2 points; Unable to carry out regular activities); ③ No evidence of infection, body temperature >38℃, ≥2 weeks; (4) No evidence of infection, night sweats >1 month
* 6. ECOG performance status of 0, 1, or 2
* 7. The main organ functions met the following criteria within 7 days before treatment: Blood routine examination criteria: platelet ≥30×10^9/L; Biochemical tests should meet the following criteria: Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase AST≤2.5*ULN; Creatinine clearance rate ≥ 30mL /min; Cardiac Doppler ultrasonography: Left ventricular ejection fraction (LVEF)≥ the lower limit of normal (50%).
* 8. Both men and women of reproductive age agreed to use reliable contraception throughout the study period and for up to four weeks after the end of treatment
* 9. Life expectancy ≥ 6 months
* 10. Patients voluntarily participated in the study and signed informed consent

Exclusion Criteria:

* 1. Have been diagnosed or treated for malignancies other than CLL (including active CNS lymphoma) within the past year
* 2. Clinical evidence suggests that Richter's transformation occurs
* 3. Non-lymphoma-related liver and kidney function impairment: ALT > 3 times the upper limit of normal value, AST > 3 times the upper limit of normal value, TBIL > 2 times the upper limit of normal value, serum creatinine clearance <30ml/min
* 4. Other serious medical conditions, such as uncontrolled diabetes, gastric ulcers, and other serious heart and lung diseases, may affect this study. The right to make judgments belongs to the researcher
* 5. Diagnosed human immunodeficiency virus (HIV) infection or active hepatitis B virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics.
* (Note: Active HBV infection was defined as a.HBV DNA quantification ≥2000 IU/ mL; b. ALT≥2 times normal upper limit; c. To exclude hepatitis caused by other causes, such as the disease itself or drugs, the three conditions must be met simultaneously. Patients with active HBV infection at initial diagnosis and non-active HBV infection after anti-HBV treatment can be included in this study on the premise of adequate anti-HBV treatment.)
* 6. Clinical manifestations of central nervous dysfunction or CNS invasion
* 7. Patients who have had major surgery (excluding lymph node biopsy) within the past 14 days or who are expected to require major surgery as part of their treatment
* 8.Unable to swallow capsules or malabsorption syndrome, disease that significantly affects gastrointestinal function, previous gastrectomy or small bowel resection, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* 9. Requires ongoing treatment with any medication which is a strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitor or strong CYP3A inducer
* 10. Females who are currently pregnant or breastfeeding, or at a childbearing age who are not using contraception
* 11. Clinically significant cardiovascular abnormalities (NYHA classification: III/IV) (Annex 3), patients with myocardial infarction, malignant arrhythmia (including QTC≥480ms), unsatisfactory blood pressure control with antihypertensive drugs (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg), and uncontrolled angina pectoris within 6 months before enrollment
* 12. Persistent uncontrolled bleeding
* 13. A history of life-threatening haemorrhage, especially from irreversible causes
* 14. High doses of several anticoagulants are required and cannot be stopped for a short time
* 15. evere allergy to the active ingredient or any excipients of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-03-22 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-11-29 (Estimated)

PRIMARY OUTCOMES:
MRD negative rate of CR patients | up to the end of 16 cycles of treatment (each cycle is 28 days)
  The negative MRD rate of patients with CR at the end of 16 cycles of treatment

SECONDARY OUTCOMES:
overall response rate(ORR) | up to the end of 16 cycles of treatment (each cycle is 28 days)
  Defined as the proportion of patients whose BICR was assessed for CR, CRi, or PR according to IWCLL 2018 criteria at or before initiation of subsequent antitumor therapy.
Complete response (CR) | up to the end of 16 cycles of treatment (each cycle is 28 days)
  Defined as the percentage of subjects who achieved CR after treatment in the conformance population and the intentionality treatment population.
Duration of tumor remission(DOR) | up to 5 years
  Defined as the time interval between the first documented remission of disease and the first documented evidence of PD for patients in the intentional-treatment population (ITT). Exit with no progress or no recorded time of disease progression, with the date of the last examination as the end date.
time to next treatment(TTNT) | up to 5 years
  Patients in the treatment-intentionality population (ITT) were defined from the beginning of first-line treatment to the beginning of back-line treatment or the time of death.
Progress-free survival(PFS) | up to 5 years
  the time from treatment initiation until disease progression or death, If there was no progress at the time of withdrawal or the time of disease progression was not recorded, the end date was the date of the last examination.
The time at which the median MRD turned positive | up to 5 years
  It was defined as the time for the median peripheral and/or bone marrow MRD to become positive in patients with CR/CRi and MRD negative in bone marrow and peripheral blood after the 16th cycle of treatment.
overall survival | up to 5 years
  Defined as the time interval from enrollment to death for patients in the treatment-intentionality population (ITT). If the patient remains alive or if it is not known whether the patient is alive or dead, the date of death will be adopted at the most recent point in time when the patient is known to be alive.
Safety of treatment regimens | up to 5 years
  Defined as treatment-related toxicity

OTHER OUTCOMES:
biological factors | up to 5 years
  To explore the effects of different biological factors on treatment response, MRD negative and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Principal Investigator — Blood disease hospital, Chinese Academic Medical School
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davids MS, Brander DM, Kim HT, Tyekucheva S, Bsat J, Savell A, Hellman JM, Bazemore J, Francoeur K, Alencar A, Shune L, Omaira M, Jacobson CA, Armand P, Ng S, Crombie J, LaCasce AS, Arnason J, Hochberg EP, Takvorian RW, Abramson JS, Fisher DC, Brown JR; Blood Cancer Research Partnership of the Leukemia & Lymphoma Society. Ibrutinib plus fludarabine, cyclophosphamide, and rituximab as initial treatment for younger patients with chronic lymphocytic leukaemia: a single-arm, multicentre, phase 2 trial. Lancet Haematol. 2019 Aug;6(8):e419-e428. doi: 10.1016/S2352-3026(19)30104-8. Epub 2019 Jun 14. PMID 31208944
- [Result] Bottcher S, Ritgen M, Fischer K, Stilgenbauer S, Busch RM, Fingerle-Rowson G, Fink AM, Buhler A, Zenz T, Wenger MK, Mendila M, Wendtner CM, Eichhorst BF, Dohner H, Hallek MJ, Kneba M. Minimal residual disease quantification is an independent predictor of progression-free and overall survival in chronic lymphocytic leukemia: a multivariate analysis from the randomized GCLLSG CLL8 trial. J Clin Oncol. 2012 Mar 20;30(9):980-8. doi: 10.1200/JCO.2011.36.9348. Epub 2012 Feb 13. PMID 22331940